CLINICAL TRIAL: NCT03236818
Title: Raising the Bars in the Treatment of Pulmonary Arterial Hypertension: Goal Oriented Strategy to Preserve Ejection Fraction Trial
Brief Title: Goal Oriented Strategy to Preserve Ejection Fraction Trial
Acronym: GOSPEL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, A. Vonk Noordegraaf, Clinical Professor, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL41878.029.13
Record Dates: First submitted 2013-03-18; First posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary arterial hypertension; right ventricle; MRI; medical combination therapy
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Sildenafil Citrate; Tadalafil; Bosentan; macitentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Upfront combination therapy (Other): Combination of an ERA and PDE-5I (Sildenafil, Tadalafil, Bosentan, Macitentan)
  Interventions: Drug: ERA and PDE-5I (Sildenafil, Tadalafil, Bosentan, Macitentan)

INTERVENTIONS:
Drug: ERA and PDE-5I (Sildenafil, Tadalafil, Bosentan, Macitentan) — Combination of an ERA and PDE-5I (Sildenafil, Tadalafil, Bosentan, Macitentan)

SUMMARY:
In this prospective long term feasibility study we examine whether a goal oriented therapeutic strategy that is able to preserve right ventricular function will result in improved clinical outcome in patients with pulmonary arterial hypertension. We hypothesize that right ventricular function can only be preserved when early and aggressive medical combination therapy not only reduces pulmonary vascular resistance but also pulmonary pressures.

DETAILED DESCRIPTION:
Rationale:

The current strategy in patients with pulmonary arterial hypertension (PAH)is to improve exercise capacity which can be achieved by decreasing pulmonary vascular resistance (PVR) and subsequently increasing cardiac output (CO). Despite this load reduction, a substantial proportion of patients show progressive right ventricular (RV) dysfunction leading to clinical worsening and death. A possible explanation is that current therapies show a relatively modest reduction in PVR, leaving mean pulmonary artery pressure (mPAP) unchanged. As a consequence RV work, defined as the product of CO and mPAP increases, contributing to progressive RV dysfunction.

Hypothesis:

A goal oriented therapeutic strategy that is able to preserve RV function will result in improved clinical outcome. RV function can only be preserved when early and aggressive combination therapy not only reduces PVR but also mPAP.

Study questions:

1. Will a goal oriented strategy to preserve/improve RV function, measured by right ventricular ejection fraction (RVEF) be effective?
2. Does early and aggressive combination therapy result in improved RV function and survival during long term follow-up?
3. Does a strategy to preserve RVEF also translate into improvements of other clinically meaningful parameters?
4. Can RVEF be replaced by more simple measures?
5. Will a goal oriented strategy to improve RVEF also lead to improvement of myocardial performances and coupling of the RV to its load?

Study design and study population:

In this prospective longitudinal feasibility study, thirty newly diagnosed idiopathic or heritable PAH patients with New York Heart Association (NYHA) functional class II or III will be included. Maintenance/improvement of RVEF will be our primary outcome parameter and therefore cardiac magnetic resonance imaging (CMR) will be performed at baseline and at 4, 8 , 12 and 24 months of follow-up. Six-minute walk testing (6MWT), quality of life questionnaires and blood sampling (NT-proBNP) will be performed at similar follow-up intervals. In addition, right heart catheterization (RHC) will be performed at baseline, after 4, 12 and 24 months of follow-up.

NYHA II patients will start with single agent medical treatment whereas patients with NYHA III will start on combination therapy (2 treatments). In case of a stable/improved RVEF during each follow-up measurement (defined as no decrease in RVEF >3% compared to previous measurement), the treatment strategy will remain unchanged. In case of decreased RVEF >3%, additional medical therapy will be added. Our hypothesis will prove to be correct when the additional medical treatment result in improved RVEF during the subsequent follow-up measurement.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic or heritable pulmonary arterial hypertension
* New York Heart Association (NYHA) functional class II or III

Exclusion Criteria:

* Other causes of pulmonary arterial hypertension (i.e. collagen vascular disease, congenital heart disease, chrono-thromboembolic pulmonary hypertension, pulmonary venous hypertension, left heart failure, hypoxemic lung disease)
* Pulmonary arterial hypertension targeted therapies before study inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-05; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Change in right ventricular ejection fraction | 4,12, 24 months of follow-up
  The primary endpoint will be change in right ventricular ejection fraction (RVEF) during 2 years of follow-up.

SECONDARY OUTCOMES:
pulmonary vascular resistance | 4,12, 24 months of follow-up
  Change in pulmonary vascular resistance
mPAP | 4,12, 24 months of follow-up
  Change in mPAP
Cardiac output in L/min (Thermodilution method) | 4,8, 12, 24 months of follow-up
  Change in cardiac output
Exercise capacity | 4,8, 12, 24 months of follow-up
  Change in exercise capacity
New York Heart Association functional class | 4,8, 12, 24 months of follow-up
  Change in New York Heart Association functional class

OTHER OUTCOMES:
NT-proBNP | 4,8, 12, 24 months of follow-up
  Change in NT-proBNP
Quality of Life by SF-36 questionnaire | 4,8, 12, 24 months of follow-up
  Change in Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Anton Vonk Noordegraaf, MD, PhD, Principal Investigator — VU University Medical Center, department of pulmonary diseases
Locations (1):
- VU University Medical Center, dept Pulmonary diseases, Amsterdam, Netherlands